CLINICAL TRIAL: NCT03108651
Title: Mobile Motivational Messages for Change (3M4Chan) Intervention in TMU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Shabbir Syed Abdul, Assistant Professor & Health IT Consultant, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N201702069
Record Dates: First submitted 2017-03-24; First posted 2017-04-11 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Explore Successful Method to Quit Smoking

STUDY DESIGN:
Intervention Model Description: Intervention study with two parallel arms.
Who Masked: Participant
Masking Description: Researchers do not disclose about App and messages to control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case (Active Comparator): Motivational message will be administrated.
  Interventions: Other: Case
- Control (No Intervention): Motivational message will not be administrated.

INTERVENTIONS:
Other: Case — Motivational message will be administrated.
  Arms: Case

SUMMARY:
About 100 (50 from TMU Hospital and 50 from Wellcome Clinic) current smokers will be recruited who contact smoke cession clinics in teaching hospitals of Taipei Medical University (TMU) and Wellcome Clinic. They will be randomly assigned either to Usual Care (UC) or Usual Care plus 3M4Chan Intervention group (IG). A randomized comparative effectiveness trial will be conducted. Patient will enroll from September 2017 to May 2018. In UC group, the physician provides a brief advice to quit during first consultation, a quit plan template, and medication prescription (Varenicline, Bupropion, Champix, Nicotinell TTS20) as decided by the physician. IG group includes UC plus a mobile App that is programmed to push tailored messages for health concern and readiness to quit, tips for sustaining abstinence, use of interactive self-assessments, helpful cessation information. This group of smokers will benefit from tailored cessation interventions with integrated body weight management elements that take into consideration the prevailing local and cultural influences on diet and levels of physical activity. IG will be continued even after stopping of the UC.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or older and approach smoke cessation clinic at TMU hospital
* Have an Android mobile phone
* Able to read Traditional Chinese
* Willing to participate in all study components
* Willing to be followed-up for 6 months
* Smoked at least once every month in the last two years
* Current smoker

Exclusion Criteria:

* • Below 20 years on the day of enrolment

  * Not willing to participate in the study
  * Those who do not have Android mobile phone or unable to read Mandarin
  * Not willing to share medical information from EHR
  * Subjects who develop adverse effects related to the pharmacological treatment included in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Smoking cessation rate at two months | Up to 2 months
  Smoking cessation rate will be measured as the ratio of the total number of patients who relapsed with total number of patients in their group. Patients will be considered to have relapsed if they fail at least one of their urine cotinine and carbon monoxide tests.
Smoking cessation rate at four months | Up to 4 months
  Smoking cessation rate will be measured as the ratio of the total number of patients who relapsed with total number of patients in their group. Patients will be considered to have relapsed if they fail at least one of their urine cotinine and carbon monoxide tests.
Smoking cessation rate at six months | Up to 6 months
  Smoking cessation rate will be measured as the ratio of the total number of patients who relapsed with total number of patients in their group. Patients will be considered to have relapsed if they fail at least one of their urine cotinine and carbon monoxide tests.

SECONDARY OUTCOMES:
User engagement at an individual level | Up to 6 months
  Engagement at individual level will be assessed based on the rate of read messages by the patients. This is calculated as the quotient between the messages the patients have read, and the total number of messages the system has sent to the patients. This metric will be assessed throughout the observation until its end.
Engagement at aggregated level - Mobile application rolling retention | Up to 6 months
  The percentage of users still active N days after installation. This is a ratio of the number of users whose last day of activity is past day N to the number of users who could have been active on day N. This metric will be assessed throughout the observation until its end.
Engagement at aggregated level - Mobile application session length distribution | Up to 6 months
  The session length is defined as the length of time between the start of the application event and the end of the application event. The session length determines the engagement as it is relevant to know how much time patients spend in the app per session. This metric will be assessed throughout the observation until its end.
Engagement at aggregated level - Mobile application session frequency | Up to 6 months
  The session frequency is a measure of how often each unique patient used the app within a given time interval. This metric will be assessed throughout the observation until its end.
Engagement at aggregated level - Mobile application sessions per user | Up to 6 months
  A session is one use of the mobile application by a patient. This begins when the application is launched and ends when the application is terminated. This metric will be assessed throughout the observation until its end.
Engagement at aggregated level - Mobile application return rate | Up to 6 months
  Return rate measures the percentage of patients who return to the app on a specific time after installation. It is measured by cohort group - that is, based on when patients first opened the app. It is calculated as the ratio of the number of users active on a given period to the size of the cohort. This metric will be assessed throughout the observation until its end.
User quitting attempts | Up to 6 months
  Number of quitting attempts per patient, including the frequency of the quitting attempts.
User app behavior | Up to 6 months
  It will be measured as the time spent per app section.
User satisfaction with messages | At 6 months after enrolment.
  Patients' answers to a satisfaction questionnaire that will be handed to them at the end of the study.
User message ratings | Up to 6 months
  User's votes for each message in a 5 star scale.
User lifestyle feedback | At enrollment and at 6 months after enrollment
  Comparison of changes in user lifestyle (at baseline and after 6 months) through the combined questionnaire EQ-5D-5L.
User lifestyle feedback | At enrollment and at 6 months after enrollment
  Comparison of changes in user lifestyle (at baseline and after 6 months) through the combined questionnaire IPAQ for physical activity.
User lifestyle feedback | At enrollment and at 6 months after enrollment
  Comparison of changes in user lifestyle (at baseline and after 6 months) through the combined questionnaires SF-36.
Physical activity | Up to 6 months
  The physical activity would be measured as the total time (minutes) of activity per user, retrieved by GoogleFit in the app.

CONTACTS AND LOCATIONS:
Locations (1):
- Syed Abdul Shabbir, Taipei, Taiwan

REFERENCES:
- [Derived] Hors-Fraile S, Malwade S, Spachos D, Fernandez-Luque L, Su CT, Jeng WL, Syed-Abdul S, Bamidis P, Li YJ. A recommender system to quit smoking with mobile motivational messages: study protocol for a randomized controlled trial. Trials. 2018 Nov 9;19(1):618. doi: 10.1186/s13063-018-3000-1. PMID 30413176